CLINICAL TRIAL: NCT06307899
Title: Comparison of Immediate Effects of Different Stretching Methods for Pectoralis Minor Muscle on Scapula Position, Pectoralis Minor Muscle Length and Scapular Muscle Activation in Individuals With Shoulder Protraction
Brief Title: Immediate Effects of Different Stretching Methods for Pectoralis Minor Muscle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Tuğçe Çoban, Research Assistant, Gazi University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: E-77082166-302.08.01-639069
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Rounded Shoulder Posture
Keywords: Pectoralis Minor; Stretching; Muscle Activation
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Unilateral Corner Stretching
  Interventions: Other: Unilateral Corner Stretch
- Group 2 (Experimental): Manual Stretching
  Interventions: Other: Manual Stretching
- Group 3 (Experimental): PNF Stretching
  Interventions: Other: PNF Stretching

INTERVENTIONS:
Other: Unilateral Corner Stretch — Individuals will be positioned in a standing position with the elbow in 90° flexion and the shoulder in 90° abduction, placing the palm on a flat surface. For stretching, individuals will be asked to increase shoulder horizontal abduction by rotating the trunk anteriorly and contralaterally. The position will be maintained for 30 seconds and will be repeated 4 times with a 30-second rest between repetitions.
  Arms: Group 1
Other: Manual Stretching — Individuals will be positioned supine with the shoulder in 90º abduction and external rotation and the elbow in 90º flexion. Stretching will be applied by the physiotherapist from just distal to the elbow in the direction of horizontal abduction of the shoulder. The position will be maintained for 30 seconds and will be repeated 4 times with a 30-second rest between repetitions.
  Arms: Group 2
Other: PNF Stretching — Individuals will be in a sitting position with their hands clasped behind the head. The PM muscle will be stretched in the direction of horizontal abduction by placing the physiotherapist's hands anterior to the elbows. Passive stretching will be continued for 10 seconds, followed by 6 seconds of maximum voluntary isometric contraction of the PM muscle. The procedure will be repeated four times with 30 seconds of rest.
  Arms: Group 3

SUMMARY:
The aim of our study is to compare the effects of different stretching methods for the pectoralis minor (PM) muscle on scapula position, PM muscle length and scapular muscle activation in individuals with shoulder protraction. Unilateral corner stretching, manual stretching and proprioceptive neuromuscular facilitation (PNF) stretching methods will be applied randomly, 2 days apart, to volunteer individuals who agree to participate in our study. Three different stretching methods (unilateral corner stretching, manual stretching and PNF stretching) will be applied to individuals randomly, 48 hours apart, and PM length, PM index, scapula upward rotation and EMG values will be recorded by a blind evaluator before and after the stretching application.

DETAILED DESCRIPTION:
Our study will include individuals who volunteer to participate in the study, and informed consent will be obtained from the individuals. Shoulder protraction will be determined according to the measurement result of the distance between the posterolateral side of the acromion and the bed in the supine position of the individual. If the distance is 2.6 centimeters or more, it will be recorded as shoulder protraction posture. PM length, PM index, upward rotation angle of the scapula at 0°, 45°, 90° and 135° abduction, electromyographic (EMG) muscle activation of the upper trapezius, middle trapezius, lower trapezius and serratus anterior muscles will be evaluated by a blind evaluator before and after the stretching methods. Unilateral corner stretching, manual stretching and proprioceptive neuromuscular facilitation (PNF) stretching methods will be applied randomly, 48 hours apart. The order of Unilateral Corner Stretching, Manual Stretching and PNF Stretching methods to be applied to individuals will be assigned with the simple allocation using random allocation. SPSS (Statistical Package for Social Sciences) version 22.0 will be used to evaluate the data obtained from the study and create tables. The Shapiro-Wilk test will be used to determine the distribution of the data. Descriptive statistics of numerical variables with normal distribution will be indicated by X ± SD, descriptive statistics of numerical variables without normal distribution will be indicated by median and (IQR), descriptive statistics of categorical variables will be indicated by frequency and percentage (%). Paired Sample T test will be used for intra-group comparison of normally distributed data and Wilcoxon test will be used for intra-group comparison of non-normally distributed data. The one-way repeated measures analysis of variance (ANOVA) will be performed to compare the three groups. The statistical significance level will be set at p<0.05 and a post-hoc multiple comparisons test with Bonferroni correction will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Having a shoulder protraction posture
* Not having had a shoulder surgery before
* Agreeing to participate in the study

Exclusion Criteria:

* Cervical or shoulder pain
* Adhesive capsulitis
* Thoracic outlet syndrome
* Shoulder instability
* Shoulder surgery history
* Numbness or tingling in the upper extremity

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-07-03 (Estimated); Study Completion 2024-09-04 (Estimated)

PRIMARY OUTCOMES:
Pectoralis Minor Length | Baseline
  To measure the length of the pectoralis minor muscle, the distance between the caudal corner of the 4th rib and the inferomedial face of the coracoid process will be recorded with a tape measure.
Pectoralis Minor Length | Immediately after intervention
  To measure the length of the pectoralis minor muscle, the distance between the caudal corner of the 4th rib and the inferomedial face of the coracoid process will be recorded with a tape measure.
Pectoralis Minor Index | Baseline
  PM index will be recorded by calculating the ratio of the pectoralis minor length to the individual's height multiplied by 100.
Pectoralis Minor Index | Immediately after intervention
  PM index will be recorded by calculating the ratio of the pectoralis minor length to the individual's height multiplied by 100.
Scapula Upward Rotation Measurement | Baseline
  Individuals' scapula upward rotation measurement will be evaluated with an inclinometer in the resting position, 45º, 90º and 135º shoulder abduction positions. Three measurements will be taken with a 30-second rest interval and the average value will be calculated.
Scapula Upward Rotation Measurement | Immediately after intervention
  Individuals' scapula upward rotation measurement will be evaluated with an inclinometer in the resting position, 45º, 90º and 135º shoulder abduction positions. Three measurements will be taken with a 30-second rest interval and the average value will be calculated.
EMG Analysis | Baseline
  Individuals' upper trapezius, middle trapezius, lower trapezius and serratus anterior muscle activations will be evaluated using superficial EMG. Measurements will be taken from the dominant side.
EMG Analysis | Immediately after intervention
  Individuals' upper trapezius, middle trapezius, lower trapezius and serratus anterior muscle activations will be evaluated using superficial EMG. Measurements will be taken from the dominant side.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Başar, PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borstad JD, Ludewig PM. Comparison of three stretches for the pectoralis minor muscle. J Shoulder Elbow Surg. 2006 May-Jun;15(3):324-30. doi: 10.1016/j.jse.2005.08.011. PMID 16679233
- [Background] Rosa DP, Borstad JD, Pogetti LS, Camargo PR. Effects of a stretching protocol for the pectoralis minor on muscle length, function, and scapular kinematics in individuals with and without shoulder pain. J Hand Ther. 2017 Jan-Mar;30(1):20-29. doi: 10.1016/j.jht.2016.06.006. Epub 2016 Oct 18. PMID 27769843
- [Background] Williams JG, Laudner KG, McLoda T. The acute effects of two passive stretch maneuvers on pectoralis minor length and scapular kinematics among collegiate swimmers. Int J Sports Phys Ther. 2013 Feb;8(1):25-33. PMID 23439770